CLINICAL TRIAL: NCT00972049
Title: A Phase I, Single-centre, Randomised, Double-blind, Placebo-controlled Parallel Group Study to Assess the Safety, Tolerability and Pharmacokinetics After Oral Single Ascending Doses of AZD2516 in Young and Elderly Japanese Healthy Subjects
Brief Title: Study to Assess Safety, Tolerability and Pharmacokinetics After Single Dose of AZD2516 to Japanese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: AstraZeneca, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D2080C00004
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2010-03-04 (Estimated); Status verified 2010-03

CONDITIONS: Healthy
Keywords: safety; tolerability; AZD2516; pain; Japanese
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Capsule administered once orally
  Interventions: Drug: AZD2516
- 2 (Placebo Comparator): Capsule administered once orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD2516 — Capsule administered once orally. Specific dose depends on dose panel.
  Arms: 1
Drug: Placebo — Capsule administered once orally
  Arms: 2

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of AZD2516 following administration of a single dose to Japanese healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Weight between 45 to 100 kg and a body mass index (BMI) between 19 to 28 kg/m2
* Japanese males aged between 20 to 45 years old (young) and Japanese males or females aged between 65 to 80 years old (elderly)

Exclusion Criteria:

* History of previous or ongoing somatic or psychiatric disease/condition
* Abnormalities in ECG that may interfere with interpretation of data.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of AZD2516 in Japanese healthy subjects by assessment of adverse events, vital signs, laboratory variables and ECG | Assessments taken at visit 1 (enrolment), defined time points pre dose and post dose during visit 2 (residential period): days -1 through to day 3 and follow up visit 3

SECONDARY OUTCOMES:
Investigate the single ascending dose pharmacokinetics of AZD2516 in Japanese subjects | Blood sampling at defined timepoints during residential period and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Anders Neijber, MD, PhD, Study Director — AstraZeneca R&D Södertälje; Shunji Matsuki, MD, PhD, Principal Investigator — Kyusyu Clinical Phramacology Research Clinic
Locations (1):
- Research Site, Fukuoka, Japan